CLINICAL TRIAL: NCT03094988
Title: COgnitive and Physical Exercise (COPE) Prehabilitation to Improve Outcomes in Surgical Patients: A Pilot Feasibility Study
Brief Title: COgnitive and Physical Exercise (COPE) Prehabilitation Pilot Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Christopher Hughes, Associate Professor of Anesthesiology, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 161802
Record Dates: First submitted 2017-03-06; First posted 2017-03-29 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Cognitive Impairment; Physical Impairment; Postoperative Complications
MeSH Terms: conditions — Cognitive Dysfunction; Postoperative Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Other): The active attention control group will receive a binder with information about personal health including sleep hygiene, nutritional changes, and stress reduction. In addition, they will participate in a control version of the cognitive training program. They will receive weekly phone calls by cognitive and physical therapy teams to address issues with any aspects of the program.
  Interventions: Other: Active attention control
- Cognitive and physical prehabilitation (Experimental): The intervention group will receive the prehabilitation program consisting of a guided progressive program of home-based aerobic and resistance training exercise, which will be adapted based on kinesiologist recommendation for each individual and the individual's perceived exertion. In addition, they will have access to the full cognitive training program. They will receive weekly phone calls by cognitive and physical therapy teams to address issues with any aspects of the program.
  Interventions: Behavioral: Cognitive and physical prehabilitation

INTERVENTIONS:
Behavioral: Cognitive and physical prehabilitation — Participants engage in cognitive and physical training daily for approximately 2-4 weeks prior to surgery.
  Arms: Cognitive and physical prehabilitation
Other: Active attention control — Participants will be provided with personal health educational materials and access to the control version of cognitive training program.
  Arms: Control

SUMMARY:
Cognitive and functional impairment are debilitating problems for survivors of major surgery. Efforts to modify medical treatments to prevent such impairment are ongoing and may yet yield significant benefits. An area in need of study is whether building patients' cognitive and physical reserve through a prescribed program of cognitive and physical exercise before the physiological insult (a prehabilitation effort) can improve long-term outcomes. Prehabilitation efforts before surgery thus far have focused on preemptive physical therapy to improve post-surgical functional outcomes. No work, however, has been done to attenuate the cognitive decline commonly seen after surgical illness by exercising the brain before the surgical insult. Cognitive prehabilitation is a novel therapeutic approach that applies well-understood techniques derived from brain plasticity research. Our approach is bolstered by data that demonstrate that cognitive training programs are effective and have a very high likelihood of fostering improvement in patient outcomes across a range of populations. It is not yet known if these programs can improve cognitive reserve, allowing patients' minds to better manage the acute stress of surgery and hospitalization. The primary aim of this pilot study is to evaluate the feasibility of cognitive and physical prehabilitation training in adult patients undergoing major non-cardiac surgery who are at risk for postoperative cognitive and functional decline. The secondary aim is to study the effects of cognitive and physical prehabilitation training on cognitive abilities, functional status, and quality of life after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adults undergoing major surgery with the likelihood of prolonged hospitalization or critical illness among the following surgical services: general surgery, surgical oncology, otolaryngology, hepatobiliary, thoracic, and vascular surgery

Exclusion Criteria:

* Blind, deaf, or unable to speak English, as these conditions would preclude our ability to perform the proposed cognitive and physical program
* Pregnancy
* Prisoners
* Severe frailty or physical impairment that prohibits participation in prehabilitation program
* Patients with documented dementia or cognitive impairment that precludes ability to self-consent for surgery and study participation
* Less than 2 weeks from scheduled surgery
* Patients without home internet access

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Participation log and diary | From date of randomization to surgery, approximately 4 weeks
  Proportion of eligible days that patients performed the cognitive and physical prehabilitation program, duration of time per day patients spent on each program

SECONDARY OUTCOMES:
Cognitive assessment | Approximately 1 month after surgery at the post-surgical clinic follow-up
  NIH toolbox cognitive battery
Instrumental activities of daily living | Approximately 1 month after surgery at the post-surgical clinic follow-up
  FAQ questionnaire
Activities of daily living | Approximately 1 month after surgery at the post-surgical clinic follow-up
  ADL questionnaire
Functional exercise capacity | Approximately 1 month after surgery at the post-surgical clinic follow-up
  2 min walk test
Muscle strength | Approximately 1 month after surgery at the post-surgical clinic follow-up
  Hand grip strength
Pulmonary function | Approximately 1 month after surgery at the post-surgical clinic follow-up
  Incentive spirometry
Acute brain dysfunction | During hospital stay after surgery, for up to 2 weeks
  Delirium
Discharge location | From time of surgery until time of discharge or death, whichever came first, assessed up to 30 days
  Determination of location where patient was discharged from hospital to, including home, nursing facility, rehab
Pain levels | During hospital stay, for up to 2 weeks, and approximately 1 month after surgery at the post-surgical clinic follow-up
  CPOT
Pain levels | During hospital stay, for up to 2 weeks, and approximately 1 month after surgery at the post-surgical clinic follow-up
  NRS
Hospital length of stay | From time of surgery until time of discharge or death, whichever came first, assessed up to 30 days
  Duration of hospital stay

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Result] Rengel KF, Mehdiratta N, Vanston SW, Archer KR, Jackson JC, Thompson JL, Pandharipande PP, Hughes CG. A randomised pilot trial of combined cognitive and physical exercise prehabilitation to improve outcomes in surgical patients. Br J Anaesth. 2021 Feb;126(2):e55-e57. doi: 10.1016/j.bja.2020.11.004. Epub 2020 Dec 13. No abstract available. PMID 33317805